CLINICAL TRIAL: NCT00453934
Title: h-Patch vs. Pen or Needle and Syringe as Insulin Administration Device in Type 1 or 2 Diabetes Patients Using MDI: Patient Preference and Glycemic Control After Switch in an Open-Label, Randomized Cross-Over Study
Brief Title: Patient Preference of h-Patch vs. Pen or Needle/Syringe as Insulin Administration Device
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Endpoint no longer deemed meaningful
Sponsor: Valeritas, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: V4001
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2007-12-06 (Estimated); Status verified 2007-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Diabetes; Type 1 Diabetes; Type 2 Diabetes; Physiologic Insulin; Basal Insulin; Bolus Insulin; Mealtime insulin; Insulin patch; Multiple daily injections
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: h-Patch

SUMMARY:
The primary objective of this study is to compare patient preference of the h-Patch as delivery device for insulin lispro compared with either an insulin pen or needle and syringe in patients with diabetes, either Type 1 or Type 2, on stable multiple daily injection regimens. This will be assessed using an accepted preference scale.

DETAILED DESCRIPTION:
Patients with Type 1 Diabetes have an absolute deficiency in insulin production and benefit from physiologic insulin replacement, defined as administration of background and mealtime insulin. More than half of patients with Type 2 diabetes (T2DM) have less than 50% of their beta cell function at the time of diagnosis. Because of this, these patients would also benefit from the physiologic delivery of insulin. Currently, 4 or more injections per day are required to deliver the various different available insulins in a physiologic manner. Valeritas has developed the h-Patch, a device suitable to make the delivery of basal and bolus insulin effective, simple and discrete. This study will measure patient preference, glucose control and safety of the h-Patch compared with patients' previous therapy. Patients previous therapy will be multiple daily injections delivered either by pens or needle and syringe.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 1or Type 2 diabetes mellitus for at least a year
2. Stable insulin regimen for at least 3 months consisting of multiple daily injections of human regular or rapid acting insulin at meal times and long or intermediate acting insulin as basal. In this protocol multiple daily injections requires at least three injections daily.
3. Total daily insulin dose between 50 and 80 units.
4. If patient is Type 2, can be treated with metformin and/or a thiazolidinedione and/or a sulfonylurea, but other diabetes drugs including α-glucosidase inhibitors, meglitinides, pramlintide exenatide, and DPP-IV's are excluded.
5. HbA1c > 7.0% and < 9.0%.

Exclusion Criteria:

1. Recurrent major hypoglycemia or prolonged unstable blood glucose control (as judged by the Investigator).
2. Use of other diabetes drugs including α-glucosidase inhibitors, meglitinides, pramlintide, exenatide or DPP-IV inhibitors (metformin and/or a thiazolidinedione and/or a sulfonylurea are allowed).
3. Intend to use any other concomitant drug therapy (prescription or over-the-counter medications) that can affect blood glucose levels.
4. Have used systemic glucocorticoids within 1 month prior to Screening or currently on glucocorticoids.
5. Have a history of drug or alcohol abuse within 1 year prior to Screening Visit.
6. Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, or neurological disease that would, in the investigator's opinion, preclude safe participation in the study.
7. Have a history of major surgery, e.g. laparotomy, thoracotomy, open orthopedic procedure, etc. within 3 months prior to Screening Visit.
8. Evidence of significant neuropsychiatric disease.
9. Have participated in a medical, surgical, or pharmaceutical investigational new drug/device study in the last 30 days or ≤ 5 half-lives of the investigational drug, whichever is longer, prior to Screening Visit.
10. Blood donation of 500 ml or more in the last 2 months prior to Screening Visit.
11. Evidence of significant active hematological disease.
12. Acute infection with fever.
13. Hemoglobin < 10 g/dL; AST, ALT ≥ 1.5 times the upper reference limit at Screening.
14. Uncontrolled treated/untreated hypertension (systolic blood pressure > 155 mmHg and diastolic blood pressure > 90 mmHg).
15. History of proliferative retinopathy or maculopathy requiring acute treatment
16. Mental incapacity, unwillingness or language barrier precluding adequate understanding or co-operation.
17. Any condition that the Investigator and/or Sponsor feel would interfere with trial participation or evaluation of results
18. Pregnancy, breast-feeding, intention of becoming pregnant for female patients of child-bearing potential.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-05; Study Completion 2007-09 (Actual)

SECONDARY OUTCOMES:
Mean glucose using CGM. | 4 weeks
Glucose SD, MAGE, Proportion of 24 hours in euglycemic range 70-160 mg/dl, using CGM. | 4 weeks
End of Study Patient Questions | 4 weeks
Hypoglycemia | 4 weeks
Proportion of time with glucose < 70 mg/dl, from CGM. | 4 weeks
Number and type of adverse events. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Kipnes, MD, Principal Investigator — Diabetes and Glandular Research
Locations (1):
- Diabetes and Glandular Research, San Antonio, Texas, United States